CLINICAL TRIAL: NCT00915213
Title: Incidence of Fluoroquinolone Resistant Enterobacteraciae in Patients Undergoing Repeat Ultrasound Guided Prostate Biopsy
Brief Title: Incidence of Antibiotic Resistant E.Coli in Patients Undergoing Repeat Prostate Biopsy
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Copan Diagnostics, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas E. Ahlering, MD, University of California, Irvine
Other Study IDs: 2008-6418
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Bacterial Infection
Keywords: E. Coli; Prostate Biopsy
MeSH Terms: conditions — Bacterial Infections; Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Rectal Swab
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Repeat Prostate Biopsy: Men who undergo repeat prostate biopsy

SUMMARY:
The purpose of this study is to discover how often certain bacteria are found in the rectum at the time of a prostate needle biopsy to diagnose prostate cancer. Certain bacteria are of importance because they can cause serious infection. Antibiotics that urologists commonly use to prevent these bacteria from causing infection are no longer effective. Many physicians around the world are noting increased infections with antibiotic resistant bacteria. Therefore; despite treating patients who are to undergo prostate biopsy with antibiotics, certain patients are being readmitted to the hospital with a serious infection. In order to study the incidence of these particular bacteria, the best method is to culture the bacteria at the time of the biopsy. This involves one rectal culture swab just prior to needle biopsy of the prostate. Once the incidence of these bacteria is known we may take steps to prevent the serious infections that occur as a result of prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* adult males
* repeat prostate biopsy

Exclusion Criteria:

* first time prostate biopsy
* minors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men undergoing repeat prostate biopsy
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2008-10; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atreya Dash, MD, Principal Investigator — University of California, Irvine
Locations (3):
- United States (3):
  - Kaiser Permanente, Irvine, California
  - Long Beach Veteran Affairs, Long Beach, California
  - University of California, Irvine Medical Center, Orange, California